CLINICAL TRIAL: NCT03681509
Title: The Effects of the Dopamine Receptor Agonist Pramipexole on Reward and Emotion Related Information Processing in Healthy Volunteers
Brief Title: Pramipexole and Emotional Processing
Acronym: PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MS IDREC R07790
Record Dates: First submitted 2018-09-19; First posted 2018-09-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Emotions; Motivation; Reward; Dopamine
Keywords: Pramipexole
MeSH Terms: interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pramipexole (Experimental): Maximum daily dose: 1.0 mg of pramipexole salt
  Interventions: Drug: Pramipexole
- Placebo (Placebo Comparator): Lactose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pramipexole — Pramipexole
  Arms: Pramipexole
Drug: Placebo — Lactose placebo capsule
  Arms: Placebo

SUMMARY:
The dopamine agonist pramipexole has recently been suggested as a potential novel antidepressant drug. While preliminary clinical data hint at its efficacy in treating depressive symptoms, our current understanding of its impact on neurocognitive processes is relatively limited. This is in part because mechanistic studies have largely focused on the effects of single-dose treatments. However, such acute administration of dopaminergic drugs likely has different cognitive effects than the more prolonged administration that is used clinically. This study therefore aims to explore and characterise the neurocognitive effects of more prolonged pramipexole treatment. Forty healthy volunteers will be randomly allocated to 12 to 15 days of treatment with either pramipexole or placebo. Study participants as well as researchers will be blinded as to which treatment is used. Before and after treatment all participants will perform a set of psychological tasks and questionnaires evaluating reward-based learning, emotional information processing, motivational vigour and subjective experience. Furthermore, functional magnetic resonance imaging (fMRI) will be used to compare neural activity during emotion and reward processing between the two treatment groups. We hypothesises that pramipexole might enhance reward sensitivity, motivational vigour, and pleasure experience and could induce positive biases in emotional information processing.

DETAILED DESCRIPTION:
Background:

The dopamine receptor agonist pramipexole has recently been suggested as a potential novel antidepressant drug. While preliminary clinical data hint at its efficacy in treating depressive symptoms, our current understanding of its impact on neurocognitive processes is relatively limited. This is in part because, so far, mechanistic studies have largely focused on the effects of single-dose treatments. However acute administration of dopaminergic drugs likely has different cognitive effects than the more prolonged administration that is used clinically.

Aim of study:

To explore and characterise the effects of a 12 to 15 day regime of pramipexole on behavioural and neural measures of reward learning, emotional information processing, motivational invigoration, and subjective experience.

Methods:

Using a double-blind, parallel-group design, forty healthy volunteers (male and female, aged 18 to 45 years) will be randomly allocated to a 12 to 15 day regime of either pramipexole (maximum daily dose of 1.0 mg pramipexole salt) or placebo. At baseline and after 12 to 15 days of treatment, a set of previously established cognitive tasks and questionnaires tapping into reward learning, emotional information processing, motivational invigoration and subjective experience will be administered. Furthermore, at 12 to 15 days of treatment, all participants will undergo functional magnetic resonance imaging to compare neural responses to reward- and emotion-related information.

Hypotheses:

Our working hypothesis is that pramipexole will enhance reward sensitivity, motivational invigoration and hedonic experience and might positively bias emotional information processing.

Implications:

This will be the first study to broadly explore and characterise the neurocognitive effects of pramipexole administered for a clinically relevant time period. The results of the study will add to our understanding of the cognitive mechanisms through which pramipexole could exert both its beneficial as well as its adverse clinical effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age: 18 to 45 years
* Good physical and mental health
* Participant is willing and able to give informed consent for participation in the study
* Sufficient knowledge of English language to understand and complete study tasks
* Willingness to refrain from driving, cycling, or operating heavy machinery if necessary while taking part in the study
* Willingness to refrain from drinking while taking part in the study.

Exclusion Criteria:

* Current or past psychiatric disorder (e.g. depression, bipolar disorder etc.)
* First-degree relative with a diagnosis of schizophrenia-spectrum or other psychotic disorder, or bipolar disorder
* BMI not between 18 and 30
* History of unexplained hallucinations or impulse control problems (e.g. pathological gambling)
* Any severe medical condition not stabilized at the time of the experiment (e.g. cardiovascular disease, epilepsy, asthma etc.)
* Severe heart or blood vessel disease
* Postural hypotension
* Any history of seizures
* Lactose intolerance
* Any current or past physical illness that has the potential to significantly affect mental functioning (e.g. epilepsy, hypothyroidism, Parkinson's disease, multiple sclerosis etc.)
* Pregnant, or lactating woman
* Sexually active woman who does not use any medically accepted method of contraception
* Current or previous intake (last three months) of any medication that has a significant potential to affect mental functioning (e.g. benzodiazepines, antidepressants, neuroleptics etc.)
* Any intake of recreational drugs in the last 3 months (e.g. marijuana, ecstasy etc.)
* Regular alcohol consumption of more than 14 units a week or excessive alcohol consumption up to three days before the experiment
* Regular smoker (> 5 cigarettes per day)
* Excessive caffeine user (> 6 caffeinated drinks per day)
* History of recurrent rashes or history of allergic reactions to relevant substances (pramipexole treatment, placebo treatment, taste samples)
* Previous participation in a study using the same or similar tasks
* Any contraindication to magnetic resonance imaging (e.g. metallic implant, severe claustrophobia)
* Current participation in another study
* In the researcher's opinion participation in the study could be harmful or severely distressing to the participant (e.g. intolerance of side effects) or the participant is not able to follow instructions or complete study tasks

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Change in reward sensitivity on a reinforcement learning task between baseline and final day of assessment | Completed at day 12 to 15 of treatment
  Participants are shown two distinct abstract shapes and have to choose one of them. On each trial, one of the two shapes is associated with a 'win' (resulting in a small monetary gain) and one with a 'loss' (resulting in a small monetary loss). The two outcomes are independent (knowing the location of the win provides no information about the location of the loss). During the task, the information content of the outcomes is manipulated independently by varying the volatility of their occurrence (three conditions: 'win volatile, loss volatile', 'win stable, loss volatile', 'win volatile, loss stable'). Using trial and error, participants have to learn the stimulus-outcome associations and use their knowledge to maximise monetary earnings. Choices are made via button-press. Choice, choice reaction time and pupillary dilation in response to outcome presentation are recorded. By fitting a computational model, reward sensitivity is estimated.

SECONDARY OUTCOMES:
Change in performance in a facial expression recognition task | Completed at day 12 to 15 of treatment
  Participants are presented with individual pictures of facial expressions of emotions. Each presented face displays one of six basic emotions (anger, disgust, fear, happiness, sadness, or surprise). Each emotional expression is presented at different levels of intensity which have been created by combining shape and texture features of the two extremes "neutral" (0%) and "full prototypical emotion" (100%) to varying degrees. Examples of neutral facial expressions are presented as well. Participants are instructed to correctly classify each facial expression as angry, disgusted, fearful, happy, sad, surprised or neutral both as quickly and as accurately as possible. Responses are made by pushing one out of seven labelled keys on a response box. Hit rates, false alarm rates, and reaction times for correct classifications are measured separately for each emotion.
Change in performance in an emotional categorisation task | Completed at day 12 to 15 of treatment
  Participants are presented with positive and negative personality descriptors and are asked to classify the valence of each word. These words describe either extremely agreeable/positive characteristics (e.g. "cheerful", "honest", "optimistic") or extremely disagreeable/negative characteristics (e.g. "domineering", "untidy", "hostile") and are presented individually in the centre of the screen. Participants are instructed to imagine themselves overhearing someone describing them with each of the words and to indicate as quickly and accurately as possible whether they would like or dislike to be described with each of the words. Responses are made by pressing a correspondingly labelled key on a button box. Reaction times for correct classifications are measured separately for positive and negative words.
Change in performance in an emotional faces dot probe task | Completed at day 12 to 15 of treatment
  Pictures of positive and negative emotional stimuli (happy and fearful facial expressions) are presented individually together with a matched neutral stimulus (neutral face). On each trial, one stimulus is shown above and the other below a central fixation point. Subsequently, a probe appears behind one of the stimuli and participants have to correctly classify the probe as quickly and as accurately as possible. Stimuli can be masked (i.e. presented very briefly and followed by a jumbled face) or unmasked (i.e. presented for a longer period without a subsequent masking stimulus). Reaction times for correct responses are recorded and vigilance scores are calculated for masked and unmasked positive and negative stimuli by subtracting reaction time data from trials when the probe appeared in the same position as the emotional stimulus (congruent trials) from trials when the probe appeared in the opposite position to the emotional stimulus (incongruent trials).
Change in performance in an emotional recall task | Completed at day 12 to 15 of treatment
  Following a delay period after the emotional categorization task (about 15 min), emotional recall memory is assessed. Participants are asked to recall and write down as many words as possible from the emotional categorization task. Numbers of correctly and incorrectly recalled positive and negative words are measured.
Amygdala BOLD signal in response to positive and negative emotional faces | Completed at day 12 to 15 of treatment
  Participants are presented with pictures of positive and negative facial expressions of emotions during functional magnetic resonance imaging. Participants are asked to correctly identify the gender of each face. BOLD signal in the amygdala in response to positive and negative emotional stimuli is measured.
Change in performance in a probabilistic instrumental learning task | Completed at day 12 to 15 of treatment
  In each trial, participants are presented with one out of two pairs of symbols. One pair of symbols is a 'win' condition in which one symbol (the 'correct' one) has a 70% chance to win a small monetary reward and a 30% chance to win nothing, while the other symbol (the 'wrong' one) has a 30% chance to win and a 70% chance to win nothing. The other pair of symbols is a 'loss' condition in which one symbol (the 'correct' one) has a 70% chance to lose nothing and a 30% chance to lose a small monetary reward, while the other symbol (the 'wrong' one) has a 70% chance to lose and a 30% chance to lose nothing. Participants are asked to choose one symbol in each pair such that they maximise their payoff. Participants have to learn the stimulus-outcome associations by trial and error such that they consistently choose the symbol with the high-probability win and low-probability loss. Responses are made via button press. Choice, reaction time, and payoff are measured.
Change in performance in a motivational vigour task | Completed at day 12 to 15 of treatment
  On each trial, participants are asked to fixate on the center of a computer screen. Following that, they are presented with a cue that provides information about how reward will be determined in that trial. Reward is determined according to one of the following four conditions: (a) 'performance-based reward' (fastest 50% of trials rewarded), (b) 'random reward' (50% small monetary reward and 50% no reward, regardless of performance), (c) 'guaranteed reward' (a fixed small monetary reward, regardless of performance), (d) 'guaranteed absence of reward' (no reward, regardless of performance). Subsequently, a target appears on either the left or the right side of the screen and participants have to move their eyes as quickly as possible towards the target. Participants are then informed about their speed and reward for the task. Saccade velocity and pupillary dilation in response to outcome are recorded.
Subjective taste experience | Completed at day 12 to 15 of treatment
  Participants are provided with standardized samples of different taste qualities (sweet, sour, bitter, salty) at four different concentrations. Participants are asked to correctly identify the taste quality of each sample and indicate on a visual analogue perceived pleasantness and disgustingness of each sample.
Change in subjective experience of pleasure | Completed at day 12 to 15 of treatment
  Snaith-Hamilton Pleasure Scale, standard questionnaire to assess subjective experience of pleasure
BOLD signal in the ventral striatum, orbitofrontal cortex and anterior cingulate cortex in response to positive and negative outcomes in a probabilistic instrumental learning task | Completed at day 12 to 15 of treatment
  Participants perform the same probabilistic instrumental learning task mentioned above while fMRI is conducted. BOLD signal in the ventral striatum and prefrontal cortex in response to positive and negative outcomes is measured.

OTHER OUTCOMES:
Change in subjective mood and energy | Completed at day 12 to 15 of treatment
  Zersen's Befindlichkeits-Skala
Change in positive and negative affect | Completed at day 12 to 15 of treatment
  Positive and Negative Affect Schedule
Change in subjective anxiety | Completed at day 12 to 15 of treatment
  State-Trait Anxiety Inventory
Change in subclinical depressive symptoms | Completed at day 12 to 15 of treatment
  Beck Depression Inventory
Change in happiness levels | Completed at day 12 to 15 of treatment
  Oxford Happiness Questionnaire
Change in subjective experience of pleasure 2 | Completed at day 12 to 15 of treatment
  Temporal Experience of Pleasure Scale
Assessment of drug-induced side effects | Completed at day 12 to 15 of treatment
  Side effect questionnaire
Change in impulsive compulsive symptoms | Completed at day 12 to 15 of treatment
  Adapted Questionnaire for Impulsive Compulsive Disorders in Parkinson's Disease Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael Browning, MB.BS, Principal Investigator — University of Oxford
Locations (1):
- Dept of Psychiatry, University of Oxford, Oxford, Oxfordshire, United Kingdom